CLINICAL TRIAL: NCT04530435
Title: PEP Flute-selfcare to Prevent Respiratory Deterioration and Hospitalization Among COVID-19 Patients: a Randomized Trial
Brief Title: PEP Flute-selfcare in COVID-19
Acronym: PEP-CoV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Berit Lilienthal Heitmann, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0211-00023B
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2; Respiratory symptoms; Positive expiratory pressure; Positive expiratory pressure flute; Airway clearance techniques
MeSH Terms: conditions — COVID-19; Signs and Symptoms, Respiratory

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomised, controlled, open-label trial with two parallel groups and a primary endpoint of CAT-score after 30 days of intervention.
  Randomization lists will be computer-generated using an appropriate statistical software and based upon permuted random blocks. The allocation ratio will be 1:1 stratified for the following baseline conditions:
  * Sex
  * Age (≥60 and <60 years)
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to treatment allocation where possible. This is of outmost importance, and participants are requested not to disclose their allocation when outcomes are assessed. To test the blinding efficacy, the outcome assessors are asked what treatment strategy they think a patient has received after assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The participants will be handed three airway resistances equivalent to a resistance of 10-20 cm H2O alongside one PEP flute. Two videos will guide the participants in use of the PEP flute; one with instructions of the rationale and how to use the flute, including how to choose the suitable resistance and one video, which gives instructions of hygienic maintenance.
  Participants in the intervention group will be advised to continue use of their PEP flute in the active intervention period of 30 days or at least if they still have respiratory symptoms. They will receive daily text-messages to prompt their reporting and to use the PEP flute according to instructions.
  Interventions: Device: PEP flute
- Control group (No Intervention): The participants in the control group will receive daily text-messages to prompt their reporting of CAT-scores. To avoid attrition of the trial due to early recovery of symptoms, the project manager will call the participants by phone at day 15 to ask them about their present condition (i.e. CAT-score) and address potential concerns of continued participation of the trial. Otherwise, they will only receive usual care.

INTERVENTIONS:
Device: PEP flute — Participants are advised to use a PEP flute at least three times daily at an appropriate resistance. Ideally, each session consists of 15 breaths (for approximately 1 minute) repeated twice at an upright position.
  Arms: Treatment group

SUMMARY:
Most research on the coronavirus SARS-CoV-2 and COVID-19 disease relate to screening measures, development of vaccines and optimising treatment of hospitalised patients. It is likely that this pandemic will be ongoing for several years until a high level of immunity is reached in the population or a vaccine has been developed. Thus, there is a need of measures to help the SARS-CoV-2 infected individual at home to overcome the course of disease with less symptoms and strain. A Positive Expiratory Pressure (PEP) flute is feasible for home use and it is possible that regular use of PEP flute may prevent the progression of respiratory symptoms in non-hospitalized individuals with COVID-19 disease.

The primary objective of the study is to examine the effect of PEP flute use among SARS-CoV-2 infected, non-hospitalized patients on self-reported change in COPD Assessment Test (CAT) score during 30 days of follow-up.

The secondary objectives are to compare the development in hospitalization rates and use of antibiotics in the intervention group and the control group during the follow-up period.

DETAILED DESCRIPTION:
It is hypothesized that the PEP flute has positive effects on SARS-CoV-2 infected individual's self-reported respiratory symptoms such as dyspnoea, coughing and perceived mucus clearance through beneficial effects on lung function and airway clearance. Furthermore, the investigators expect a lower rate of hospitalization and use of antibiotics in the intervention group as compared to the control group.

Finally, potential subgroup effects by gender, age, comorbidity and BMI at study entry will be explored for all outcomes.

Based upon a sample size estimation the investigators assess that inclusion of 200 participants in each intervention arm will be an adequate number. Based on the present testing strategy and COVID-19 incidence, current expectations are that two months should be enough to recruit 400 patients. The investigators will allow for recruitment to the end of December 2020, but will terminate enrolment at n = 400.

Link to detailed protocol paper will be added once published.

ELIGIBILITY:
Inclusion Criteria:

* Positive SARS-CoV-2
* Symptoms of SARS-CoV-2 infection e.g. fever, cough and shortness of breath.
* Access to use a smartphone
* Can reply to a questionnaire (sent on email, text messages or via telephone interview) in Danish
* Given informed consent

Exclusion Criteria:

* Age < 18 years.
* Any condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation, such as psychiatric disorders.
* Hospitalised patients or citizens living in nursing homes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Self-reported CAT-score (COPD Assessment Test) | Day 30.
  CAT-scores will be measured using a telephone administered questionnaire. The CAT-score is validated to evaluate symptoms in COPD patients. Eight items covers symptoms of cough, sputum, chest pain, dyspnoea, activities of daily living at home, feeling safe at home despite symptoms (modified for the present study from feeling safe at leaving home despite symptoms), sleep quality and vigour. The eight items sum up to a range of 0-40 with higher scores indicating more respiratory impairment. Although validated for COPD-use, the CAT-scale is considered useful in the present study because several of the items (dyspnoea, cough, fatigue, sputum and pleuritic chest pain) previously have been used as outcome variables in pneumonia studies. The outcome assessment can be taken within + 1 week for the scheduled visit.

SECONDARY OUTCOMES:
Hospital admissions | Up to day 30, 90 and 180.
  Will be obtained from the Danish National Patient Registry, from which also data of comorbidity will be retrieved.
Use of antibiotics | Up to day 30, 90 and 180.
  Will be obtained from the Danish National Prescription Registry.
Self-reported CAT-score (COPD Assessment Test) | Day 90, Day 180.
  CAT-scores will be measured using a telephone or email-administered questionnaire. The outcome assessment can be taken within + 1 week for the scheduled visit.

OTHER OUTCOMES:
Serious Adverse Events | During treatment, up to 30 days.
  Assessed by Common Terminology Criteria for Adverse Event (CTCAE).
General and respiratory symptoms | Day 30, 90, Day 180.
  Measured according to the COVIDmeter from Statens Serum Institut using a telephone or email-administered questionnaire. The outcome assessment can be taken within + 1 week for the scheduled visit.

CONTACTS AND LOCATIONS:
Overall Officials: Berit L. Heitmann, Professor, Ph.D, Principal Investigator — Research Unit for Dietary Studies at the Parker Institute, Bispebjerg and Frederiksberg Hospitals, Denmark
Locations (1):
- Research Unit for Dietary Studies at the Parker Institute, Bispebjerg and Frederiksberg Hospitals, Frederiksberg, Denmark

REFERENCES:
- [Derived] Mollerup A, Henriksen M, Larsen SC, Bennetzen AS, Simonsen MK, Kofod LM, Knudsen JD, Nielsen XC, Weis N, Heitmann BL. Effect of PEP flute self-care versus usual care in early covid-19: non-drug, open label, randomised controlled trial in a Danish community setting. BMJ. 2021 Nov 24;375:e066952. doi: 10.1136/bmj-2021-066952. PMID 34819329
- [Derived] Mollerup A, Larsen SC, Bennetzen AS, Henriksen M, Simonsen MK, Weis N, Kofod LM, Heitmann BL. PEP-CoV protocol: a PEP flute-self-care randomised controlled trial to prevent respiratory deterioration and hospitalisation in early COVID-19. BMJ Open. 2021 Jun 30;11(6):e050582. doi: 10.1136/bmjopen-2021-050582. PMID 34193503